CLINICAL TRIAL: NCT02502448
Title: Impact of Acute Normovolemic Hemodilution on Whole Blood Coagulation Profile During Post-cardiopulmonary Bypass in Cardiac Surgery: Rotational Thromboelastometry Study
Brief Title: Acute Normovolemic Hemodilution on ROTEM in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KUH1160030
Record Dates: First submitted 2015-03-03; First posted 2015-07-20 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Mitral Regurgitation; Mitral Stenosis; Tricuspid Regurgitation
Keywords: rotational thromboelastometry; cardiac surgery; acute normovolemic hemodilution
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis; Tricuspid Valve Insufficiency | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): patients undergoing cardiac surgery supposed not to get aucte normovolemic hemodilution (ANH) before CPB
- Acute normovolemic hemodilution group (Active Comparator): patients undergoing cardiac surgery supposed to get aucte normovolemic hemodilution (ANH) before CPB
  Interventions: Procedure: Acute normovolemic hemodilution (ANH); Drug: hydroxyethyl starch (HES 130/0.6)

INTERVENTIONS:
Procedure: Acute normovolemic hemodilution (ANH) — applying acute normovolemic hemodilution (ANH) by using HES 130/0.4 of 5 ml/kg before the initiation of cardiopulmonary bypass
  Arms: Acute normovolemic hemodilution group
Drug: hydroxyethyl starch (HES 130/0.6)
  Arms: Acute normovolemic hemodilution group

SUMMARY:
Impact of acute normovolemic hemodilution (ANH) using hydroxyethyl starch before initiating cardiopulmonary bypass (CPB) on whole blood viscoelastic profile after CPB has not been well established.

Patients undergoing cardiac surgery employing moderate hypothermic CPB (n=40) are randomly allocated into one of two groups: in Group-ANH(n=20), ANH is applied by using a balanced hydroxyethyl starch (HES 130/0.6); and in Group-C, ANH is not applied.

After weaning from CPB, intergroup differences of INTEM, EXTEM, FIBTEM and APTEM profiles are analyzed.

As a primary outcome, inter-group difference between maxiaml clot firmness of EXTEM will be determined at 10 min after ANH in Group-ANH and that at control.

DETAILED DESCRIPTION:
Background: Impact of acute normovolemic hemodilution (ANH) using hydroxyethyl starch before initiating cardiopulmonary bypass (CPB) on whole blood viscoelastic profile after CPB has not been well established.

Method: Patients undergoing cardiac surgery employing moderate hypothermic CPB (n=40) are randomly allocated into one of two groups: in Group-ANH(n=20), ANH is applied by using a balanced hydroxyethyl starch (HES 130/0.6); and in Group-C ANH is not applied.

Intergroup differences of INTEM, EXTEM, FIBTEM and APTEM profiles are analyzed. after anesthesia induction (control) and after weaning form CPB and protamine neutralization (after-CPB) in both groups. In Group-ANH, those are determined after ANH (after-ANH).

As a primary outcome, inter-group difference between maxiaml clot firmness of EXTEM is determined at 10 min after ANH in Group-ANH and that at control.

As secondary outcomes, intergroup differences of Hematocrit (Hct), Na+, K+, HCO3-, Ca2+, osmolarity, s-Cr are determined Intergroup difference of data at T2 are performed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery with cardiopulmonary bypass who signed written informed consent

Exclusion Criteria:

* preoperative renal failure requiring reran replacement therapy
* preoperative liver disease
* preoperative low cardiac output (EF < 50%)
* Preoperative IABP application, Atrial fibrillation, Pacemaker,
* contraindication for applying TEE
* intraoperative withdrawal

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximal clot firmness of EXTEM | 10 min after completion of acute normovolemic hemodilution (ANH)
  Maxiaml clot firmess (MCF) of EXTEM of rotational thromboleastometry

SECONDARY OUTCOMES:
Clot formation time of EXTEM | 10 min after completion of acute normovolemic hemodilution
  Clot formation time of EXTEM of rotational thromboleastometry
A10 of FIBTEM | 10 min after completion of acute normovolemic hemodilution
  A10 of FIBTEM of rotational thromboelastometry

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea